CLINICAL TRIAL: NCT03352206
Title: Community Studies to Monitor the Impact of Triple Drug Therapy Relative to Double Drug Therapy on Lymphatic Filariasis Infection Indicators
Brief Title: Prevalence Studies After Triple Drug Therapy for Lymphatic Filariasis
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Case Western Reserve University (Other); Ministere de la Sante Publique et de la Population, Haiti (Unknown); Indonesia University (Other); Papua New Guinea Institute for Medical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201710040
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Lymphatic Filariases
Keywords: Mass drug administration; Effectiveness
MeSH Terms: conditions — Elephantiasis, Filarial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2-Drug Treated Communities: Communities who were treated with diethylcarbamazine and albendazole (DA) mass drug administration during the safety study entitled "Community Based Safety Study of 2-drug (DA) versus 3-drug (IDA) Therapy for Lymphatic Filariasis."
  Interventions: Drug: 2 drug dose - DA
- 3-Drug Treated Communities: Communities who were treated with ivermectin, diethylcarbamazine and albendazole (IDA) mass drug administration during the safety study entitled "Community Based Safety Study of 2-drug (DA) versus 3-drug (IDA) Therapy for Lymphatic Filariasis."
  Interventions: Drug: 3 drug dose - IDA

INTERVENTIONS:
Drug: 2 drug dose - DA — Lymphatic Filariasis Mass Drug Administration (MDA) with the currently used standard of care combination drug therapy of diethylcarbamazine and albendazole (DA)
  Other Names: DA
  Groups: 2-Drug Treated Communities
Drug: 3 drug dose - IDA — Lymphatic Filariasis Mass Drug Administration (MDA) with triple drug therapy of ivermectin, diethylcarbamazine, and albendazole (IDA)
  Other Names: IDA
  Groups: 3-Drug Treated Communities

SUMMARY:
This study will assess the impact of 2-drug (DA) or 3-drug (IDA) regimens on lymphatic filariasis infection parameters in communities. Parameters measured will include: circulating filarial antigenemia (CFA) assessed with the Filariasis Test Strip (FTS), antifilarial antibodies tested with plasma and microfilaremia (assessed by night blood smears and microscopy).

DETAILED DESCRIPTION:
Results from clinical trials in Papua New Guinea and Cote d'Ivoire have shown that a single dose of three drugs (ivermectin, diethylcarbamazine, and albendazole [IDA]) was superior to standard two drug therapy (diethylcarbamazine and albendazole [DA]) in clearing W. bancrofti microfilaremia (MF) (King et al. unpublished data).1 Recently, large safety studies that treated more than 23,000 participants across four countries were conducted to determine if IDA was safe for use in mass drug administration (MDA) (DOLF Project, unpublished data). Currently, there is no information about what community indicators of infection look like following shorter IDA programs. It is possible that current WHO guidelines for stopping MDA need to be modified for MDA programs that use IDA. Observing the levels of infection indicators in a community following treatment with IDA will provide important information to the GPELF if IDA is recommended for use in MDA programs. There is an opportunity to study communities that were treated with IDA during the "Community Based Safety Study of 2-drug (Diethylcarbamazine and Albendazole) versus 3-drug (Ivermectin, Diethylcarbamazine and Albendazole) Therapy for Lymphatic Filariasis". Communities in this study were randomly assigned to receive IDA or DA treatment. A large percentage of individuals in these communities participated in the study thereby approximating a mass distribution of the treatments. By surveying these communities 12 months following their initial treatment the investigators will be able to better understand and compare the impact of MDA with IDA or DA on LF infection parameters at the level of communities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years (males and females)
* Able to provide informed consent, or parental/guardian consent for young children, and assent for older children

Exclusion Criteria:

* Unable or unwilling to provide informed consent or (for minors) lacking parental/guardian consent to participate in the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All eligible individuals who reside in the communities where the "Community Based Safety Study of 2-drug (Diethylcarbamazine and Albendazole) versus 3-drug (Ivermectin, Diethylcarbamazine and Albendazole) Therapy for Lymphatic Filariasis" was conducted.
Sampling Method: Probability Sample
Enrollment: 20092 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with circulating filarial antigenemia (CFA) as measured by the Filaria Test Strip | One sample collected about 12 months after exposure to treatment
  To assess the impact of DA vs. IDA mass drug administration in community settings participants will be tested using the filaria test strip (FTS) which detects circulating filarial antigen.
Number of participants with IgG4 antifilarial antibodies in plasma | One sample collected about 12 months after exposure to treatment
  To assess the impact of DA vs. IDA mass drug administration in community settings participant's dried blood spot specimens will be tested using a commercially available antibody test.
Number of participants with microfilaremia as measured with night blood smear testing | One sample collected about 12 months after exposure to treatment
  To assess the impact of DA vs. IDA mass drug administration in community settings participants with positive FTS will be tested for presence of microfilaria detected by thick blood smear using 60 microliters (ul) from finger prick blood collected at night.

SECONDARY OUTCOMES:
Community prevalence of microfilaremia as measured with night blood smear | One comparison about 12 months after exposure to treatment
  Community prevalence of microfilaremia will be compared between the two cohorts to identify any difference of the impact of mass drug administration with IDA or DA
Community prevalence of circulating filarial antigen as measured with filarial test strip | One comparison about 12 months after exposure to treatment
  Community prevalence of circulating filarial antigen will be compared between the two cohorts to identify any difference of the impact of mass drug administration with IDA or DA
Prevalence of STH (hookworm, ascaris, trichuris and strongyloides) as measured by Kato-katz or PCR | One comparison about 12 months after exposure to treatment
  Some sites will include stool sample collections to compare the impact of MDA with IDA or DA on soil transmitted helminth (STH) infection parameters in communities. Stool samples will be analyzed using Kath-katz method, as well as PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Weil, MD, Principal Investigator — Washington University School of Medicine
Locations (5):
- Ministry of Health and Medical Services, Suva, Fiji
- Ministere de la Sante Publique et de la Population, Port-au-Prince, Haiti
- Vector Control Research Centre, Puducherry, India
- Universitas Indonesia, Jakarta, Indonesia
- Papua New Guinea Institute for Medical Research, Madang, Papua New Guinea

IPD SHARING:
Plan to Share IPD: Yes
Datasets used for published results will be shared publically through a journal or other open source data repository so that the broader scientific community can access it. Only de-identified data will be shared publicly.

REFERENCES:
- [Background] Thomsen EK, Sanuku N, Baea M, Satofan S, Maki E, Lombore B, Schmidt MS, Siba PM, Weil GJ, Kazura JW, Fleckenstein LL, King CL. Efficacy, Safety, and Pharmacokinetics of Coadministered Diethylcarbamazine, Albendazole, and Ivermectin for Treatment of Bancroftian Filariasis. Clin Infect Dis. 2016 Feb 1;62(3):334-341. doi: 10.1093/cid/civ882. Epub 2015 Oct 20. PMID 26486704
- [Background] Hooper PJ, Chu BK, Mikhailov A, Ottesen EA, Bradley M. Assessing progress in reducing the at-risk population after 13 years of the global programme to eliminate lymphatic filariasis. PLoS Negl Trop Dis. 2014 Nov 20;8(11):e3333. doi: 10.1371/journal.pntd.0003333. eCollection 2014 Nov. PMID 25411843
- [Background] Ichimori K, King JD, Engels D, Yajima A, Mikhailov A, Lammie P, Ottesen EA. Global programme to eliminate lymphatic filariasis: the processes underlying programme success. PLoS Negl Trop Dis. 2014 Dec 11;8(12):e3328. doi: 10.1371/journal.pntd.0003328. eCollection 2014 Dec. No abstract available. PMID 25502758
- [Background] Irvine MA, Stolk WA, Smith ME, Subramanian S, Singh BK, Weil GJ, Michael E, Hollingsworth TD. Effectiveness of a triple-drug regimen for global elimination of lymphatic filariasis: a modelling study. Lancet Infect Dis. 2017 Apr;17(4):451-458. doi: 10.1016/S1473-3099(16)30467-4. Epub 2016 Dec 22. PMID 28012943
- [Background] World Health Organization. Monitoring and Epidemiological Assessment of Mass Drug Administration in Global Programme to Eliminate Lymphatic Filariasis: A Manual for National Elimination Programmes. Geneva: World Health Organization; 2011. http://www.who.int/lymphatic_filariasis/resources/9789241501484/en/. Accessed October 11, 2017.
- [Background] World Health Organization. Assessing the epidmiology of soil-transmitted helminths during a transmission assessment survey in the global programme for the elimination of lymphatic filariasis. 2015. http://apps.who.int/iris/bitstream/10665/153240/1/9789241508384_eng.pdf. Accessed October 12, 2017.
- [Derived] Laman M, Tavul L, Karl S, Kotty B, Kerry Z, Kumai S, Samuel A, Lorry L, Timinao L, Howard SC, Makita L, John L, Bieb S, Wangi J, Albert JM, Payne M, Weil GJ, Tisch DJ, Bjerum CM, Robinson LJ, King CL. Mass drug administration of ivermectin, diethylcarbamazine, plus albendazole compared with diethylcarbamazine plus albendazole for reduction of lymphatic filariasis endemicity in Papua New Guinea: a cluster-randomised trial. Lancet Infect Dis. 2022 Aug;22(8):1200-1209. doi: 10.1016/S1473-3099(22)00026-3. Epub 2022 May 6. PMID 35533701